CLINICAL TRIAL: NCT02147223
Title: Sex-dependent Effects of Flavanol Metabolism and Absorption on Vascular Status
Brief Title: Sex-dependent Effects of Flavanols on Vascular Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BRANDED
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases
Keywords: flavanols; sex-related cardiovascular effects
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Flavanol rich product A (Active Comparator): 250 mg flavanols
  Interventions: Dietary Supplement: Flavanol rich intervention; Dietary Supplement: Flavanol free intervention
- Flavanol rich product B (Active Comparator): 500 mg flavanols
  Interventions: Dietary Supplement: Flavanol rich intervention; Dietary Supplement: Flavanol free intervention
- Flavanol rich product C (Active Comparator): 750 mg flavanols
  Interventions: Dietary Supplement: Flavanol rich intervention; Dietary Supplement: Flavanol free intervention
- Flavanol free product (Placebo Comparator): flavanol free
  Interventions: Dietary Supplement: Flavanol rich intervention

INTERVENTIONS:
Dietary Supplement: Flavanol rich intervention — Flavanol intervention products (250 mg, 500 mg and 750 mg flavanols)
Dietary Supplement: Flavanol free intervention — Calorically, micro- and macronutrient matched control product free of flavanols
  Arms: Flavanol rich product A; Flavanol rich product B; Flavanol rich product C

SUMMARY:
Epidemiological studies suggest that certain foods rich in flavanols, including cocoa products, red wine, and tea, are associated with decreased cardiovascular mortality and morbidity. Dietary interventional studies have corroborated this finding and showed that flavanols can acutely and after sustained ingestion improve surrogate markers of cardiovascular risk including endothelial function. Endothelial dysfunction is the key event in the development and progression of cardiovascular disease. The aim of the study is to assess sex specific effects of cocoa flavanols on endothelial and vascular function in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy post-menopausal femal subjects (>50 years)
* healthy male subjects (>50 years)

Exclusion Criteria:

* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* CRP > 1 mg/dl
* malignant disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Absolute change of Flow-mediated Vasodilation (FMD) | 2 hours

SECONDARY OUTCOMES:
Pulse wave velocity | 2 hours
  Measured by SphygmoCor
Augmentation index | 2 hours
  Measured by SphygmoCor
Ambulatory blood pressure | 2 hours
  automatical measurements
Plasma flavanol metabolites | 2 hours
  Measured by HPLC
laboratory safety parameters | 2 hours
  blood/urine samples for safety assessment (haematology, biochemistry, and urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Ana Rodriguez Mateos, PhD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine, Düsseldorf, Germany